CLINICAL TRIAL: NCT01142141
Title: Manual Therapy in Postoperative Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Maria Teresa Pace do Amaral
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 095/2006
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer; Axillary Lymph Node Dissection; Shoulder Joint Limitation
MeSH Terms: conditions — Breast Neoplasms | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manual therapy, kinesiotherapy (Other)
  Interventions: Other: manual therapy, kinesiotherapy

INTERVENTIONS:
Other: manual therapy, kinesiotherapy

SUMMARY:
To evaluate the effectiveness of manual therapy (joint mobilization and massage) combined with kinesiotherapy in women with impaired range of motion after axillary lymph node dissection due to breast cancer regarding the recovery of shoulder range of motion and functionality of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* surgery of breast cancer at University of Campinas
* axillary lymph node dissection
* injury of shoulder range of motion

Exclusion Criteria:

* bilateral surgery
* previous radiotherapy
* bone metastasis in homolateral upper limb
* axillary web syndrome

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil